CLINICAL TRIAL: NCT01551108
Title: Parent-targeted Mobile Phone Based Intervention to Increase Physical Activity in Children (P-Mobile)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: The Coca-Cola Company (Industry)
Responsible Party: Principal Investigator, Robert Newton, Principal Investigator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PBRC 11022
Record Dates: First submitted 2012-03-08; First posted 2012-03-12 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Physical Activity
Keywords: Children; physical activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mobile phone intervention: minimal (Active Comparator): Intervention: limited behavioral strategies
  Interventions: Behavioral: Intervention: limited behavioral strategies
- Mobile phone intervention: intensive (Experimental): Intervention: advanced behavioral strategies
  Interventions: Behavioral: Intervention: advanced behavioral strategies

INTERVENTIONS:
Behavioral: Intervention: limited behavioral strategies — Parents are given access to a website, formatted for a mobile phone. The website provides parents with a target steps/day goal for their child and parents are instructed to use their mobile phone to access the study website to record their child's step count each night. Parents are also sent monthly healthy nutrition tips via text message targeting the child in order to provide these families with potentially health promoting information.
  Arms: Mobile phone intervention: minimal
Behavioral: Intervention: advanced behavioral strategies — Parents are given access to a website, formatted for a mobile phone. The website provides parents with a target steps/day goal for their child and parents are instructed to use their mobile phone to access the study website to record their child's step count each night. Parents also receive additional behavioral strategies based on the Social Cognitive Theory. The strategies are delivered through weekly articles posted on the website. Text messages are designed to prompt parents to encourage their child's physical activity, remind parents of behavioral concepts presented in the articles (article tip), and motivate parents to foster behavioral change in their child.
  Arms: Mobile phone intervention: intensive

SUMMARY:
This study is designed to determine if parents can deliver an intervention that will help increase physical activity in their children. The parents will be given the intervention through their mobile phones.

DETAILED DESCRIPTION:
Most children engage in insufficient amounts of moderate-to-vigorous physical activity. These low levels of moderate-to-vigorous physical activity are associated with adverse health consequences including increased risk for obesity, and cardiovascular and diabetes risk factors. Therefore, there is a need for studies that can increase physical activity levels in children. Mobile phones are a way to deliver behavioral interventions. Mobile phones are portable, allow for real-time data collection, and can potentially reach large numbers of people. Text messages can also be utilized to promote behavior change. Few mobile phone based interventions have specifically targeted child physical activity.

The aims of this pilot study were to determine the feasibility and efficacy of a physical activity promotion program targeting 6-10 year old children that is delivered to parents through mobile phones.

ELIGIBILITY:
Inclusion Criteria:

* Parent must own a mobile phone.
* Parent must use the text (SMS)messaging service on their mobile phone.
* Parent can access the internet on their mobile phone.

Exclusion Criteria:

* Child is 6 through 10 years old.
* Child does not engage in regular physical activity.
* Chile is physically capable of exercising.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2012-03; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Step counts | 3 Months
  Physical activity will be measured by utilizing pedometers.

SECONDARY OUTCOMES:
Waist circumference, body mass index, blood pressure | 3 Months
  Physical measurements will be assessed by waist circumference, body mass index, height, weight, percent body fat, and blood pressure. Questionnaires will assess mood and physical activity enjoyment.

CONTACTS AND LOCATIONS:
Overall Officials: Robert L. Newton, Jr., PhD, Principal Investigator — Pennington Biomedical Research Center; Timothy Church, MD,MPH,PhD, Principal Investigator — Pennington Biomedial Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Derived] Newton RL Jr, Marker AM, Allen HR, Machtmes R, Han H, Johnson WD, Schuna JM Jr, Broyles ST, Tudor-Locke C, Church TS. Parent-targeted mobile phone intervention to increase physical activity in sedentary children: randomized pilot trial. JMIR Mhealth Uhealth. 2014 Nov 10;2(4):e48. doi: 10.2196/mhealth.3420. PMID 25386899